CLINICAL TRIAL: NCT00484822
Title: Multicentric, Randomized, Controlled, Double-blind Clinical Trial to Assess Perioperative Bridging Therapy With Sodium Bemiparin vs Calcium Unfractionated Heparin in Invasive Procedures, Outpatient Surgery and Laparoscopy Surgery in Patients Receiving Long-term Oral Anticoagulant Therapy
Brief Title: Bemiparin Randomized Trial on Bridging Oral Anticoagulants in Invasive Procedures (BERTA Study)
Acronym: BERTA
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study has been halted prematurely due to a low recruitment.
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Institut de Recerca Hospital de la Santa Creu i Sant Pau, Institut de Recerca Hospital de la Santa Creu i Sant Pau
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACO-BEMI-01-2006; 2006-001862-17
Record Dates: First submitted 2007-06-08; First posted 2007-06-11 (Estimated); Last update posted 2010-02-04 (Estimated); Status verified 2010-02

CONDITIONS: Long-term Oral Anticoagulant Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Brazo 1: Bemiparina Sódica 3.500 UI/día.
  Interventions: Drug: Bemiparina Sodica
- 2 (Placebo Comparator): Brazo 2: Heparina Cálcica 10.000 UI/día.
  Interventions: Drug: Heparina Cálcica

INTERVENTIONS:
Drug: Bemiparina Sodica — 3.500 UI/día.
  Arms: 1
Drug: Heparina Cálcica — 10.000 UI/día.
  Arms: 2

SUMMARY:
Often it is necessary to temporarily discontinue OAT when surgical or other invasive procedures are required. However, there is no consensus on the optimal management in these situations, and heparin bridging therapy is the current usual practice in these situations. No large randomized, controlled clinical trials have been yet performed to evaluate the efficacy and safety of a low molecular weight heparins (LMWH) as bridging therapy.

DETAILED DESCRIPTION:
THE MAIN OBJECTIVE of this study is to evaluate the efficacy and safety of the subcutaneous administration of Bemiparin 3,500 IU, for the peri-operative procedural management of patients requiring temporary interruption of oral anticoagulation therapy (OAT).

PRIMARY EFFICACY ENDPOINT: combined incidence of arterial and venous thromboembolic events and deaths from any causes within 3 months after the invasive procedure.

PRIMARY SAFETY ENDPOINT: incidence of major bleeding within 10 days after the invasive procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over 18 years who have given their informed consent to participate in the study.
2. Patients receiving oral anticogulants during at least 3 months and who require outpatient surgery, laparoscopy surgery or invasive procedures
3. Procedures must be performed from 8 am to 15 pm.

Exclusion Criteria:

1. Patients with severe renal failure (creatinine clearance <30 ml/min) or hepatic insufficiency (AST and/or ALT>5 times the normal value established by the reference range of the local hospital laboratory).
2. Patients who have shown thromboembolic events with an appropriate INR.
3. Known hypersensitivity to LMWH, heparin or substances of porcine origin.
4. Patients with organic lesions susceptible to bleeding (e.g. active peptic ulcer, stroke, aneurysms).
5. Patients with a history of heparin-induced thrombocytopenia.
6. Patients with suspected inability/or inability to comply with treatment and/or complete the study.
7. Patients who are participating in another clinical trial or have been participated in the past 30 days.
8. Patients with antithrombin deficit and C and S protein deficit
9. Women who are pregnant or breast-feeding, or with the possibility of becoming pregnant during the study.
10. Acute bacterial endocarditis or slow endocarditis.
11. Severe arterial hypertension (systolic blood pressure over 200 mmHg and/or diastolic blood pressure over 120 mmHg).
12. Patients with antiplatelet therapy
13. Patients with mechanical cardiac valves in mitral position and body weight 90 Kg with/or bone mass index (BMI) > 30 or 50 kg
14. Patients with Starr-Edwards valves.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2007-02; Study Completion 2009-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Fontcuberta Boj Jordi, Dr., Study Chair — Fundació de Gestió Sanitaria del hospital de la Santa Creu i Sant Pau
Locations (31):
- Spain (31):
  - Hospital General de Alicante, Alicante, Alicante
  - Hospital de Torrevieja, Torrevieja, Alicante
  - Hospital Tries I Pujol, Badalona, Barcelona
  - Hospital Del Mar, Barcelona, Barcelona
  - Fundació de Gestió Sanitaria de l'Hospital de la Santa Creu i sant Pau, Barcelona, Barcelona
  - Hospital Sagrado Corazón, Barcelona, Barcelona
  - Hospital de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Mataró, Mataró, Barcelona
  - Hospital Mútua Terrassa, Terrassa, BARCELONA
  - Hospital Consorci Sanitari de Terrassa, Terrassa, Barcelona
  - Hospital Puerta Del Mar, Cadiz, Cadiz
  - Hospital Provincial de Castellón, Castellon, Castellón
  - Hospital General de Castellón, Castellon, Castellón
  - Hospital de La Plana, Villarreal, Castellón
  - Hospital Vinaroz, Vinaròs, Castellón
  - Hospital de Jerez, Jerez de la Frontera, Cádiz
  - Hospital Virgen de Las Nieves, Granada, Granada
  - Hospital Arnau de Vilanova, Lleida, Lleida
  - Hospital La Princesa, Madrid, Madrid
  - Hospital Morales Messeguer, Murcia, Murcia
  - HOSPITAL DE NAVARRA (Pamplona), Pamplona, Navarre
  - Hospital Comarcal de Valdeorras, O Barco de Valdeorras, Ourense
  - Hospital Son Dureta, Palma de Mallorca, Palma de Mallorca
  - Hospitalson Llàtzer, Palma de Mallorca, Palma de Mallorca
  - Hospital Clínica Universitaria Pamplona, Pamplona, Pamplona
  - Hospital Universitario de Salamanca, Salamanca, Salamanca
  - Hospital Joan Xxiii, Tarragona, Tarragona
  - HOSPITAL TORTOSA (Verge de la Cinta), Tortosa, Tarragona
  - Hospital de La Ribera, Alzira, Valencia
  - HOSPITAL ARNAU DE VILANOVA(Valencia), Valencia, Valencia
  - Hospital Clinico Lozano Blesa, Zaragoza, Zaragoza